CLINICAL TRIAL: NCT04613440
Title: Randomized Controlled Trial of Accessible Online Genetic Services for Cascade Testing for BRCA Mutation Carriers Versus Usual Care in a Clinic Setting
Brief Title: FaCT Trial (Facilitated Cascade Testing Trial)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Basser Research Center for BRCA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-03021615
Record Dates: First submitted 2020-10-27; First posted 2020-11-03 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: BRCA1 Mutation; BRCA2 Mutation
Keywords: Genetic Testing, Cascade, BRCA1, BRCA2
MeSH Terms: conditions — Fanconi Anemia, Complementation Group D1 | interventions — Standard of Care; Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard of care - Proband-mediated cascade testing (Other): Probands randomized to the standard of care group will be instructed to share a family letter (providing information on the familial mutation) with their FDRs and encourage FDRs to complete genetic testing.
  Interventions: Other: Family Letter (Standard of Care)
- Intervention - Facilitated cascade testing (Other): In the intervention group, a patient navigator will provide facilitated support, including an initial genetic counseling call, an email with a link to an educational video, and, for individuals who are interested in completing testing - a link to create an account for a free saliva kit and a follow-up call to discuss the results and ensure participants are connected with their primary care provider or other clinician, as appropriate.
  Interventions: Other: Educational Video; Other: Mailed Saliva Kit for Genetic Testing; Other: Telephone Counseling
- Exploratory Arm (Experimental): Probands at WCM only who do not meet eligibility criteria for randomization to the intervention and control arms will be offered enrollment in a third arm, in which they will receive the intervention in addition to the option for referral to patient advocacy/support groups including FORCE: Facing Hereditary Cancer EMPOWERED, Sharsheret, SHARE, LatinaSHARE, Oneinforty, Susan G. Komen, Any Mountain, and Genetic Support Foundation, for additional guidance. Probands enrolled in this third arm only will be asked to share the names and contact information for all first, second, and third-degree relatives with whom they have shared their genetic testing results. We estimate enrolling up to 200 subjects into this exploratory third arm (50 probands and 150 Relatives including first, second, and third-degree relatives).
  Interventions: Other: Educational Video; Other: Mailed Saliva Kit for Genetic Testing; Other: Telephone Counseling

INTERVENTIONS:
Other: Family Letter (Standard of Care) — The family letter is given to probands in the standard of care arm and provides information on the familial mutation and serves to encourage first degree relatives to complete genetic testing.
  Arms: Standard of care - Proband-mediated cascade testing
Other: Educational Video — The educational video is provided by the clinical genetic testing laboratory and explains the importance and implications of genetic testing. This educational video is shared with first degree relatives in the intervention arm
  Arms: Exploratory Arm; Intervention - Facilitated cascade testing
Other: Mailed Saliva Kit for Genetic Testing — The FDR's email will be sent to the genetic testing lab, Invitae, which will allow them to log on to the online portal, create a unique account, and order a genetic testing saliva kit free of charge. The FDR will receive the kit and instructions in the mail. The FDR will collect the saliva sample and send the sample back to the genetic testing laboratory.
  Arms: Exploratory Arm; Intervention - Facilitated cascade testing
Other: Telephone Counseling — The FDR's will be contacted and receive post genetic testing phone counseling
  Arms: Exploratory Arm; Intervention - Facilitated cascade testing

SUMMARY:
The purpose of this study is to assess an intervention that incorporates engagement strategies with a medical team navigator, an educational video and accessible genetic testing services to maximize the genetic testing and education of at-risk relatives. In this study, first degree relatives who agree to participate will either receive this intervention or standard of care. The investigators do not know if the facilitated interventional method will be more effective than the standard of care method. This research is being done because identification of patients with inherited gynecologic/breast cancer syndromes is critical to enable delivery of tailored cancer treatment and cancer prevention to both the patients and their at-risk relatives. Cascade genetic testing, defined as extending genetic testing to the family members of affected patients, results in a more precise risk assessment and initiation of appropriate cancer screening and prevention strategies. Therefore, this trial will compare the efficacy of a multicomponent facilitated intervention for first degree relatives vs. standard of care in terms of the overall proportion of first degree relatives who complete genetic testing by 6 months (primary outcome).

DETAILED DESCRIPTION:
This prospective randomized controlled trial will compare the efficacy of a multicomponent facilitated cascade testing intervention. One hundred and fifty probands with a diagnoses of a BRCA1/2 mutation will be enrolled and randomized to the intervention vs. control arms. Probands will be asked to share the names and contact information for all FDR (First Degree Relative) with whom they have shared their genetic testing results. One hundred and fifty probands will be recruited and randomized and, therefore, based on our institutional experience, the investigators anticipate on average 3 FDRs per proband, therefore up to 450 FDRs. Probands randomized to the standard of care group will be instructed to share a family letter (providing information on the familial mutation) with their FDRs and encourage FDRs to complete genetic testing. In the intervention group, a patient navigator will provide facilitated support, including an initial genetic counseling call, an email with a link to an educational video, and, for individuals who are interested in completing testing - a link to create an account for a free genetic testing saliva kit and a follow-up call to discuss the results and ensure participants are connected with their primary care provider or other clinician, as appropriate. Participating FDRs will complete quality of life assessments. FDRs found to have BRCA1/2 mutations will be followed to determine if they completed cancer risk-reducing surveillance or surgery as a result of the genetic testing results. Analyses will assess the proportion of first degree relatives who complete genetic testing by 6 months (primary outcome), as well as the proportion who engage subsequently in recommended risk-reducing behaviors by 18 months and quality of life; distributions of time between proband diagnosis and first degree relative testing; and potential covariate correlations. Probands at WCM only who do not meet eligibility criteria for randomization to the intervention and control arms will be offered enrollment in a third arm, in which they will receive the intervention in addition to the option for referral to patient advocacy/support groups including FORCE: Facing Hereditary Cancer EMPOWERED, Sharsheret, SHARE, LatinaSHARE, Oneinforty, Susan G. Komen, Any Mountain, and Genetic Support Foundation, for additional guidance. Probands enrolled in this third arm only will be asked to share the names and contact information for all first, second, and third-degree relatives with whom they have shared their genetic testing results. We estimate enrolling up to 200 subjects into this exploratory third arm (50 probands and 150 Relatives including first, second, and third-degree relatives).The combined total enrollment for the randomized probands and FDRs, and the probands and relatives (first, second, and third-degree relatives) enrolled in the third arm will total 800. To recruit patients for all arms of this study, we will identify eligible probands from any of the following sources: Genetic Counselors, Institutional Clinicians, BRCA Genetics Conferences, and by reviewing clinic schedules on weekly basis for potentially eligible patients.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older as documented in the medical record
2. Speaks and reads English or Spanish as reported by the patient
3. Patients who are currently receiving diagnostic, treatment, or follow-up care at New York Presbyterian/ Weill Cornell Medical Center, MD Anderson Cancer Center, Duke University or Columbia University.
4. Patients with a newly diagnosed BRCA mutation presenting for consultation OR patients with known BRCA mutations who have been diagnosed with a confirmed deleterious (pathogenic) variant in BRCA1, or BRCA2 within the preceding 12 months as documented in the medical record
5. BRCA1/2 mutation that is included on testing panel provided by the clinical genetic testing laboratory
6. Patients who have at least one at risk relative who meets criteria for first degree relatives

Exclusion Criteria:

1. Is unwilling or unable to provide informed consent.
2. Does not have email access.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 820 (Estimated)
Dates: Start 2021-07-21 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of genetic testing by 6 months among FDRs on each study arm | 6 months
  To compare proportion of completion of genetic testing at 6 months follow-up among first degree family relatives (referred to herein as "FDR": son, daughter, full-brother, full-sister, mother, father) of patients with a confirmed BRCA1/2 mutation (referred to as "proband") randomized to the intervention arm versus the standard of care.

SECONDARY OUTCOMES:
Proportion of first-degree relatives who subsequently engage in recommended risk-reducing behaviors by 18 months | 18 months
  To compare proportion of engagement in risk reducing behaviors by 18 month follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa K Frey, MD, MS, Principal Investigator — Weill Medical College of Cornell University
Locations (3):
- United States (3):
  - Weill Cornell Medicine, New York, New York
  - Duke University, Durham, North Carolina
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nitecki R, Moss HA, Watson CH, Urbauer DL, Melamed A, Lu KH, Lipkin SM, Offit K, Rauh-Hain JA, Frey MK. Facilitated cascade testing (FaCT): a randomized controlled trial. Int J Gynecol Cancer. 2021 May;31(5):779-783. doi: 10.1136/ijgc-2020-002118. Epub 2020 Dec 18. PMID 33443030